CLINICAL TRIAL: NCT04871633
Title: Effectiveness of Remedesvir in SARS-CoV2 Patients Presenting at Mayo Hospital Lahore
Brief Title: Effectiveness of Remedesvir in COVID-19 Patients Presenting at Mayo Hospital Lahore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 483/RC/KEMU
Record Dates: First submitted 2021-01-11; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
Keywords: Remdesvir; Sars CoV-2; Effectiveness
MeSH Terms: conditions — COVID-19 | interventions — remdesivir; Congresses as Topic; Methylprednisolone Hemisuccinate; Dexamethasone; Prednisolone; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remdesivir (Active Comparator): patients having drug Remdesivir in addition to conventional treatment according to disease grade (steroids, anticoagulants, antibiotics if needed, oxygen therapy, paracetamol, antihistamine)
  Interventions: Drug: Remdesivir; Drug: Conventional
- Conventional (Other): patients having Standard Conventional therapy only.
  Interventions: Drug: Conventional

INTERVENTIONS:
Drug: Remdesivir — Remdesivir is an intravenous (IV) loading dose of 200 mg on day 1 followed by daily IV maintenance doses of 100 mg for 5-10 days
  Other Names: Veklury
  Arms: Remdesivir
Drug: Conventional — IV Steroids Antibiotics
  Other Names: Solumedrol, dexamethasone,prednisolone, azithromycin

SUMMARY:
Currently, several drugs including Remdesivir, hydroxychloroquine, chloroquine, ritonavir+lopinavir, Tocilizumab, Arbidol and interferon are under randomised controlled trials (RCTs) for efficacy and/or safety evaluations in patients with COVID-19 in different countries. Remdesivir (GS-5734) is among these investigational drugs and some studies reported promising results. Remdesivir is a nucleotide analogue intravenous pro-drug developed by Gilead Sciences, an American biopharmaceutical company, for treatment of Ebola virus during the 2014 Ebola outbreak in Western Africa. Remdesivir shows broad-spectrum antiviral activity against many RNA viruses including SARS-CoV-2 through blocking RNA polymerase thereby terminating RNA transcription. Remdesivir was among the first treatments used in China as the outbreak emerges and it has been reported as potential treatment options for COVID-19 in the USA, China and Italy.

DETAILED DESCRIPTION:
Coronavirus diseases 2019 (COVID-19) is caused by a novel β-coronavirus which is named as SARS-CoV-2. SARS-CoV-2 shares 79% RNA sequence identity with severe acute respiratory syndrome coronavirus 2 (SARS-COV2) and 50% genomic sequence identity with Middle East respiratory syndrome coronavirus (MERS-CoV) which caused a major outbreak since 2002 and 2012 in China and Saudi Arabia, respectively. Despite global containment measures to fight the disease, the pandemic continued to rise, rapidly spread across the world, and resulting in in 10.5 million confirmed cases and 51391 deaths worldwide as of July 1st 2020. The outbreak of COVID-19 infection has a significant threat to international health, the economy, psychological stress and mental health worldwide. Yet, there are no approved vaccines or drugs to make the disease less deadly; implying that searching therapeutic options are critical issues to overcome the outbreak. Studies are strongly underway to discover rapidly drug candidates for COVID-19, and studies are looking into repurposing drugs that have been used for the treatment of other diseases.

Pakistan is badly facing this pandemic too. Up till now there are 221,896 confirmed cases with 4551 deaths with a death ratio of 2.1%. More than 3000 patients are critical.8 In Punjab, being allocated as a leading tertiary care centre for COVID-19 patients, Mayo hospital Lahore is dealing with each and every category of COVID-19 patients with variable presentations and treating those patients with different investigational drugs in keeping with other countries to find the best possible treatable drug.

US Food and Drug Administration (FDA) has issued an emergency use authorisation (EUA) of the antiviral drug remdesivir for the treatment of patients with COVID-19. Although clinical trials have showed remdesivir as a treatment option for COVID-19, results are controversial. That's why we need to conduct a trial in our part of the world too to see its effectiveness in patients presenting with Covid-19.

Remdesivir has been recently approved by CEAG (Corona Expert Advisory Group) for COVID patient is Mayo hospital. Remdesivir has never been used before in any public sector hospital in Punjab. Investigators aim to do this study in Mayo hospital Lahore to check the efficiency of this drug in COVID-19 patients in Mayo hospital Lahore

OBJECTIVE:

The objective of the study is to evaluate the effectiveness of remdesivir in patients with COVID-19 presenting to Mayo Hospital Lahore

OUTCOME AND UTILIZATION:

To date, no therapy has demonstrated efficacy for patients with COVID-19.This study will help in finding any definite role of Remdesivir in COVID -19 patients who are severely ill . Although data from several international ongoing randomized, controlled trials will soon provide more informative evidence regarding the safety and efficacy of remdesivir for COVID-19, but this needs to be evaluated in local arena too.

ELIGIBILITY:
Inclusion Criteria:

1. All Patients with confirmed COVID-19 of either gender and aged 12 years and above.
2. Patients having Severe COVID 19 Disease. Severe disease is defined as patients with an oxygen saturation (SpO2) ≤94% on room air or requiring supplemental oxygen or requiring mechanical ventilation or requiring extracorporeal membrane oxygenation (ECMO).17

   -

Exclusion Criteria:

1. Known severe allergic reaction to Remdesivir or to other antiviral drugs
2. Patients already having other treatments like tocilizumab or other antiviral drugs
3. Pregnancy or breastfeeding
4. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 times upper normal limit
5. Creatinine clearance <30ml/min
6. Low platelet count <50,000/l

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Hospital Stay | 10 days
  Duration of stay in hospital in days
Ventilation | 10 Days
  No of patients needing IPPV

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No